CLINICAL TRIAL: NCT05079555
Title: Study of the Effect of Robotic Devices on the Functional Rehabilitation of Hip Fractures in Elderly People.
Brief Title: Effect of a Robotic Platform for Hip Fracture Rehab
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Werium Assistive Solutions (Industry)
Collaborators: Albertia Servicios Sociosanitarios (Unknown)
Responsible Party: Principal Investigator, Vanina Costa, Principal Investigator, Werium Assistive Solutions
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SWalkerRehab
Record Dates: First submitted 2021-09-22; First posted 2021-10-15 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Intervention Model Description: The performance of the SWalker platform was assessed at Albertia Servicios Sociosanitarios S.A. nursing homes. Clinical validation was conducted with hip fracture patients. The control group consisted of patients who followed conventional therapy, while the intervention group consisted of patients rehabilitated using SWalker. Allocation to groups was according to the choice of the participants. All patients had the possibility to use SWalker treatment. For those patients who received conventional rehabilitation, treatment duration was up to 6 months in the most severe case. Patient follow-up was conducted in parallel with the clinical trials.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The control group consisted of patients who followed conventional therapy.
- Intervention group (Experimental): The intervention group consisted of patients rehabilitated using the robotic platform.
  Interventions: Device: Robotic rehab

INTERVENTIONS:
Device: Robotic rehab — Patients using the robotic platform SWalker
  Arms: Intervention group

SUMMARY:
Hip fracture is one of the most common traumas associated with falls in the elderly, severely affecting the patient's mobility and independence. The treatment involves hospitalization and prolonged rehabilitation periods with high costs which are associated with an increased mortality rate due to health complications. In recent years, the use of robotic applications has proven to be effective in gait rehabilitation, especially for neurological disorders. However, there is a lack of research in robotic rehabilitation focused on the hip fracture of elderly people. This study presents the validation of a novel robotic platform for hip rehabilitation called SWalker aimed at improving the rehabilitation of this condition in comparison with conventional rehabilitation.

DETAILED DESCRIPTION:
The performance of the SWalker platform was assessed at Albertia Servicios Sociosanitarios S.A. nursing homes. Clinical validation was conducted with hip fracture patients. The control group consisted of patients who followed conventional therapy, while the intervention group consisted of patients rehabilitated using SWalker. Allocation to groups was according to the choice of the participants. All patients had the possibility to use SWalker treatment. Physiological parameters, and functional assessment scales such as FAC and Tinetti were collected at the beginning and at the end of the intervention. Gait recovery and rehabilitation process indicators were also gathered. The total duration of the clinical validation was 15 months. For each patient, the total duration of treatment was between 1 week and 1 month with the robotic platform. For those patients who received conventional rehabilitation, treatment duration was up to 6 months in the most severe case. Patient follow-up was conducted in parallel with the clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Patients who, after recently having undergone a hip fracture surgery, needed subsequent rehabilitation to restore autonomous ambulation
* patients over 65 years of age

Exclusion Criteria:

* patients who have undergone a hip fracture surgery more than 5 months ago
* patients who have already received other types of hip fracture rehabilitation therapies
* patients with advanced and limiting neurological and cognitive impairment

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-04-15 (Actual)

PRIMARY OUTCOMES:
effectiveness of rehabilitation | through study completion, an average of 3 months
  Number of physiotherapy sessions
Degree of gait recovery | through study completion, an average of 3 months
  time to recovery of autonomous walking to perform their daily functional tasks (days)

CONTACTS AND LOCATIONS:
Locations (1):
- Albertia Servicios Sociosanitarios, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No